CLINICAL TRIAL: NCT02311725
Title: Narrative Intervention to Disseminate ACT for Depression in Primary Care
Brief Title: Storytelling Video Intervention for Depressed Primary Care Patients - Pilot Trial
Acronym: sTVi-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lisa Uebelacker, Co-PI, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sTVi-2; R34MH103568 (NIH)
Record Dates: First submitted 2014-12-03; First posted 2014-12-08 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2022-06

CONDITIONS: Major Depressive Disorder
Keywords: narrative communication; depression; antidepressant augmentation; primary care
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- aTAU + sTVi (Experimental): Antidepressant Treatment as Usual (aTAU): All participants will receive antidepressant treatment as usual provided by their primary care doctor during the study.
  Storytelling Video Intervention (sTVi): We will develop a series of 4 videos, each episode approximately 30 minutes long, which will illustrate the key principles of Acceptance and Commitment Therapy.
  In addition, we will develop an accompanying "personal journal" for participants that includes a brief self-help guide which encourages participants to write about what they learned in the videos and how they will take similar steps in their own lives to cope with depression.
  Interventions: Behavioral: aTAU + sTVi
- aTAU + Attention Control Videos (Active Comparator): Antidepressant Treatment as Usual (aTAU): All participants will receive antidepressant treatment as usual provided by their primary care doctor during the study.
  Attention Control Videos: Control participants will view videos about general mental health and well-being. Specifically, we plan to give participants 4 30-minute videos on topics including nutrition, stress reduction, movement and recreation, and becoming an educated patient. The series comes with an accompanying course guidebook. We will provide videos on the same schedule as sTVi.
  Interventions: Behavioral: aTAU + Attention Control Videos

INTERVENTIONS:
Behavioral: aTAU + sTVi — Antidepressant treatment as usual provided by participants' primary care physician plus narrative communication, video-based intervention for improving depression in primary care patients.
  Arms: aTAU + sTVi
Behavioral: aTAU + Attention Control Videos — Antidepressant treatment as usual provided by participants' primary care physician plus videos about general mental health and well-being on the same dose and frequency as the experimental intervention.
  Arms: aTAU + Attention Control Videos

SUMMARY:
The overall aim of this program of research is to refine and test a newly developed storytelling video intervention (sTVi) for depressed primary care patients.

The purpose of the proposed project is to establish the feasibility, acceptability, and preliminary effects of the intervention for an eventual large-scale randomized clinical trial which would test the efficacy of sTVi in comparison to a control condition.

To achieve the specific aims, the investigators will conduct a pilot randomized clinical trial (n = 40), with two treatment arms: antidepressant treatment as usual (aTAU) + sTVI vs aTAU + attention control videos.

DETAILED DESCRIPTION:
The public health impact of existing treatments for major depression is limited by our ability to disseminate those treatments. There is a particular need to find innovative ways to disseminate key principles of empirically supported psychotherapy in primary care settings. Narrative communication is an alternative way to disseminate psychotherapy behavior change principles. Narrative communication refers to "storytelling" -real people talking about their struggles and successful ways of coping. An advantage of narrative communication is that it can be easily distributed (by video) and may reach people who do not have access to other technologies or who experience barriers to traditional psychotherapy. We propose that key principles of a type of cognitive-behavioral therapy (Acceptance and Commitment Therapy, or ACT) can be readily disseminated through a video storytelling intervention. Together with a video production firm with a record of working in healthcare and developing documentary-style videos, we will produce a storytelling video intervention (sTVi).

Our specific aim is to conduct a pilot randomized controlled trial (n = 40) with depressed primary care patients who will receive either antidepressant treatment as usual (aTAU) + sTVi vs aTAU + attention control videos. Assessments will occur at baseline, 4 (post-treatment) and 12 weeks (follow-up). We will examine feasibility and acceptability of sTVi (e.g., uptake and completion of sTVi, engagement with videos, and understanding of key ACT principles), the attention control videos, and this research design. We will examine treatment differences (within relevant confidence intervals) on outcomes (e.g., depression severity). We will examine change in potential mechanisms, i.e., ACT-consistent coping strategies derived from key ACT principles.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-5 criteria for current or lifetime major depressive disorder.
2. No Lifetime diagnosis of bipolar disorder, schizophrenia, or chronic psychotic condition.
3. No current hazardous illicit drug or alcohol use.
4. No suicidal ideation or behavior requiring immediate attention.
5. Depression symptom severity: a Quick Inventory of Depressive Symptoms (QIDS) score >11.
6. Taking an antidepressant medication for at least 6 weeks; prescribed by their primary care provider.
7. Not in psychotherapy during the study period.
8. Have a PCP at our enrollment site.
9. If pregnant, less than 24 weeks gestation.
10. English speaking.
11. Aged 18 or older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Clinician Rating (QIDS-C) | 4 weeks

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire-8 (CSQ-8) | 4 weeks
Acceptance and Action Questionnaire-II (AAQ-II) | 4 weeks
WHO-Quality of Life-BREF (WHO-QOL-BREF) | 4 weeks
WHO-Disability Assessment Schedule-II (WHO-DAS-II) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Uebelacker, PhD, Principal Investigator — Butler Hospital/Brown University; Brandon Gaudiano, PhD, Principal Investigator — Butler Hospital/Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaudiano BA, Davis CH, Miller IW, Uebelacker L. Pilot randomized controlled trial of a video self-help intervention for depression based on acceptance and commitment therapy: Feasibility and acceptability. Clin Psychol Psychother. 2020 May;27(3):396-407. doi: 10.1002/cpp.2436. Epub 2020 Feb 28. PMID 32087610
- See also: Pilot randomized controlled trial of a video self-help intervention for depression based on acceptance and commitment therapy: Feasibility and acceptability — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7322697/